CLINICAL TRIAL: NCT06385847
Title: Cross-Over Trial to Assess The Patient Preference for Goserelin Microsphere Versus Goserelin Implant in Patients With Prostate Cancer
Brief Title: To Assess The Patient Preference for Goserelin Microsphere Versus Goserelin Implant in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Wang Xuegang, Associate chief physician, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GOMIMP
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, cross-over phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zo-LY (Other): Arm Zo-LY: Zoladex 3.6 mg (s.c.)/4W ✖ 2 cycles, followed by LY01005 3.6 mg (i.m.)/4W ✖ 2 cycles
  Interventions: Drug: Zoladex; Drug: LY01005
- LY-Zo (Other): Arm LY-Zo: LY01005 3.6 mg (i.m.)/4W ✖ 2 cycles, followed by Zoladex 3.6 mg (s.c.)/4W ✖ 2 cycles
  Interventions: Drug: Zoladex; Drug: LY01005

INTERVENTIONS:
Drug: Zoladex — Patients received 3.6 mg subcutaneous Zoladex
Drug: LY01005 — Patients received 3.6 mg intramuscular LY01005

SUMMARY:
The GOMIMP will be a Prospective, Randomized, Cross-over Trial to Explore the Patient Preference for Goserelin Microsphere (Zoladex®) Versus Goserelin Implant (LY01005) in Patients of Prostate Cancer

DETAILED DESCRIPTION:
Androgen Deprivation Therapy (ADT) is an important systemic therapy for prostate cancer, which plays a vital role in the treatment of various stages of prostate cancer. Gonadotropin-releasing hormone (GnRH) agonists are the most commonly used ADT treatment，including leuprolide, goserelin, and triptorelin. The goserelin implant (Zoladex®) 3.6 mg is administered subcutaneously every 28 days into the anterior abdominal wall using a pre-filled syringe with a 16G needle (outer diameter 1.6 mm), while the Goserelin microsphere (LY01005) 3.6 mg is administered every 28 days by intramuscular injection using a 21G injection needle (outer diameter 0.8 mm). Phase III study (NCT04563936) have confirmed the similar efficacy and safety between the two drugs, but patient preference for both are unknown.

The objective of this study was to explore the patient preference for goserelin microsphere versus goserelin implant in patients of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients older than 18 years
2. Histologically confirmed prostate adenocarcinoma
3. Suitable for ADT treatment
4. ECOG≤2
5. Prior treatment without GnRH agonists
6. Expected survival >1 year
7. Good compliance
8. Adequate organ or bone marrow function as evidenced by:

   * Hemoglobin >/= 10 g/dL
   * Absolute neutrophil count >/=1.5 x 109/L,
   * Platelet count >/=100 x 109/L,
   * AST/SGOT and/or ALT/SGPT </=1.5 x ULN;
   * Total bilirubin </=1.5 x ULN,
   * Serum creatinine </=1.5 x ULN. If creatinine 1.0 - 1.5 xULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded

Exclusion Criteria:

1. Prior treatment with Zoladex, LY01005 or other GnRH agonists, while GnRH agonists for < 6 months and discontinued for more than 6 months were allowed
2. Diagnosed or suspected hormone-resistant prostate cancer, hypophysectomy, adrenalectomy, or pituitary lesions
3. A history of cardiovascular events, uncontrolled hypertension, gastrointestinal disease that interferes with treatment absorption, active viral hepatitis, or human immunodeficiency infection (HIV) within the past 6 months
4. Any medical conditions that the investigators believe make the patient ineligible to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient preference | Assessed up 16 weeks after randomization
  Patient preference (assessed by a single question) between Zoladex and LY01005 after completion of the second period of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China